CLINICAL TRIAL: NCT05350293
Title: Evaluation of Two Different Types of Abutments on Post-prosthesis Bone Resorption: A Randomized Controlled Clinical and Radiological Trial
Brief Title: Evaluation of the Abutment Type Following Oral Implants in Terms of the Surrounding Bone Height
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-08-2022
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Missing Teeth
Keywords: dental implant; 3D printed abutment; molded abutment
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molded abutment (Active Comparator): A plastic abutment that is provided by the implant manufacturer will be used. This abutment will be modified using wax, and then it will be dismantled, wedged, and poured using a Ni-Cr mixture. A plastic abutment that the implant manufacturer provides will be used. This abutment will be modified using wax, and then it will be dismantled, wedged, and poured using a Ni-Cr mixture.
  Interventions: Other: Molded abutment
- 3D printed abutment (Experimental): The customised abutment will be made using a laser printer with a Cr-Co mixture after being designed using a special computer program.
  Interventions: Other: 3D printed abutment

INTERVENTIONS:
Other: Molded abutment — The waxed plastic abutment will dismantle, wedged, and poured using a Ni-Cr mixture then it will be trimmed to make it ready to make the permanent restoration over it.
  The prostheses will be cemented above the abutment using dual-cure resin cement then the final restoration (crown and abutment) will be fixed using a screw-retained manner.
  Arms: Molded abutment
Other: 3D printed abutment — A marker or Scan body appropriate for the type of implant will be placed on the laboratory implant substitute, a digital scan of the marker will be done in the lab, and the scanned image will be transferred to a computer design software where the prosthesis is designed, In the printing phase, the final prosthesis will be manufactured using a stepwise metal powder supply and a laser fusion process. Making the abutment ready to make the permanent restoration over it. The prostheses will be cemented above the abutment using dual-cure resin cement then the final restoration (crown and abutment) will be fixed using a screw-retained manner.
  Arms: 3D printed abutment

SUMMARY:
Compare two different types of abutments (molded abutments and computer-designed 3D printed abutments) in terms of the amount of bone loss, and depth of periodontal pockets around the implant during different periods.

DETAILED DESCRIPTION:
In the past few years, the number of research conducted on the designs of abutments and materials has increased. Often, the restoration is done over the implant using standard abutments that the implant company prefabricated, but due to the problems facing the dentist from the occurrence of bone absorption, an increase in the depth of the pocket after restoration, other types of abutment design methods have been introduced as needed (molded abutment made by lost wax technique and computer-designed abutment made using a 3D laser printer), those customised abutments were made special for each patient depending on their conditions.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age is greater than 20 years and younger than 50
* Good oral health
* Absence of systemic diseases that may affect the healing of surrounding tissues, such as diabetes.

Exclusion Criteria:

* The presence of non-functional habits such as stridor
* Acute or acute periodontitis, previous loss of implants
* Poor general health conditions
* Previous radiotherapy in the head and neck area
* Mental incompetence
* Orthodontic treatment

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Change in the crestal bone height | T1:3 months after cementation, T2: 6 months after cementation, T3: 1 year after cementation
  It Is the loss of bone that occurred around the dental implant neck after fixing the final prosthesis (abutment and crown).
  A periapical radiograph is going to be taken using a digital intra-oral sensor with a special holder in a parallel way, to measure the changes that occurred at the level of the bone around the implant depending on MBLS concept taking two referring points from the neck of the abutment to the first match of the bone with the abutment using special programs on computer (Photoshop) during different periods.

SECONDARY OUTCOMES:
Change in the depth of periodontal pockets | T1: direct after cementation, T2:3 months after cementation, T3: 6 months after cementation, T4: 1 year after cementation
  Periodontal pockets are spaces surrounding the implant under the gum line. The pocket around the implant will be measured by using special plastic probe slides between the implant and gum to measure the depth of the periodontal pocket, and the changes in the depth of pockets will be noted and register after fixing the final prosthesis (abutment and crown), during different periods.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Anas Almodalal, DDS,MSc, Principal Investigator — Department of fixed prosthodontics , Damascus University, Syria; Mohammad Luai Morad, DDS,MSc,PhD, Study Director — Department of fixed prosthodontics , Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbin T, Veloso DV, Del Rio Silva L, Borges GA, Presotto AGC, Barao VAR, Mesquita MF. 3D metal printing in dentistry: An in vitro biomechanical comparative study of two additive manufacturing technologies for full-arch implant-supported prostheses. J Mech Behav Biomed Mater. 2020 Aug;108:103821. doi: 10.1016/j.jmbbm.2020.103821. Epub 2020 Apr 27. PMID 32469723
- [Background] Bae S, Hong MH, Lee H, Lee CH, Hong M, Lee J, Lee DH. Reliability of Metal 3D Printing with Respect to the Marginal Fit of Fixed Dental Prostheses: A Systematic Review and Meta-Analysis. Materials (Basel). 2020 Oct 26;13(21):4781. doi: 10.3390/ma13214781. PMID 33114737
- [Background] Jang Y, Sim JY, Park JK, Kim WC, Kim HY, Kim JH. Accuracy of 3-unit fixed dental prostheses fabricated on 3D-printed casts. J Prosthet Dent. 2020 Jan;123(1):135-142. doi: 10.1016/j.prosdent.2018.11.004. Epub 2019 Apr 23. PMID 31027960
- [Background] Ramalho I, Witek L, Coelho PG, Bergamo E, Pegoraro LF, Bonfante EA. Influence of Abutment Fabrication Method on 3D Fit at the Implant-Abutment Connection. Int J Prosthodont. 2020 Nov/Dec;33(6):641-647. doi: 10.11607/ijp.6574. PMID 33284906
- [Background] Chou WT, Chuang CC, Wang YB, Chiu HC. Comparison of the internal fit of metal crowns fabricated by traditional casting, computer numerical control milling, and three-dimensional printing. PLoS One. 2021 Sep 16;16(9):e0257158. doi: 10.1371/journal.pone.0257158. eCollection 2021. PMID 34529710